CLINICAL TRIAL: NCT03232099
Title: Evaluation of Red Wine Effects Upon Gut Flora and Plasma Levels of Trimethylamine-N-oxide (TMAO) in Patients With Established Atherosclerotic Disease
Brief Title: Red Wine Effects Upon Gut Flora and Plasma Levels of Trimethylamine-N-oxide (TMAO) - WineFlora Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); IBRAVIN (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 57379216.0.0000.0068; 2015/212606 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2017-06-20; First posted 2017-07-27 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2017-05

CONDITIONS: Trimethylamine-N-oxide; Gut Microbiota; Effects of Red Wine; Atherosclerosis
Keywords: trimethylamine-N-oxide; TMAO; Gut Microbiota; Gut Flora; Atherosclerosis; Wine; Red Wine
MeSH Terms: conditions — Atherosclerosis | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Forty two men with established atherosclerotic disease will be studied:after a 2 week washout period, each subject receives both treatments, intervention and control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Red Wine group (RW) (Experimental): After a two weeks washout period,in the intervening period with red wine, patients will receive 250 mL / day of red wine per Day, 5 days a week, for 3 weeks.
  Interventions: Dietary Supplement: Red Wine consumption
- Abstemious (Active Comparator): After a two weeks washout period,in the Abstemious period, patients should not consume any kind of alcohol beverages, for 3 weeks
  Interventions: Other: Period without alcohol consumption

INTERVENTIONS:
Dietary Supplement: Red Wine consumption — After a two weeks washout period,in the intervening period with red wine, patients will receive 250 mL / day of red wine per Day, 5 days a week, for 3 weeks.
  Arms: Red Wine group (RW)
Other: Period without alcohol consumption — After a two weeks washout period,in the Abstemious period, patients should not consume any kind of alcohol beverages, for 3 weeks
  Other Names: Abstain Period
  Arms: Abstemious

SUMMARY:
Recent evidence indicates that Trimethylamine-N-oxide (TMAO) is a pro-atherosclerotic, phosphatidylcholine-dependent metabolite of diet and intestinal flora. Food substrates derive from carnitine and phosphatidylcholine (lecithin), present mainly in eggs, red meat, liver and pork. The intestinal flora pattern that favors the formation of TMAO is very similar to that which predisposes to insulin resistance and obesity: a high proportion between phylum Firmicutes over Bacteroidetes. The intestinal microbiota is sensitive and variable; the use of prebiotics and probiotics can change the relationship between Firmicutes/Bacteroidetes phyla. Red wine (RW), for its composition with polyphenols and possible bactericidal role, may play a role in the intestinal flora modification and could promote proliferation of beneficial bacteria. However, the influence of RW on TMAO is not known. This is the hypothesis to be tested in this trial. METHODS: This is a prospective, crossover, randomized, controlled trial with patients from Heart Institute (InCor), FMUSP and volunteers recruited through press releases. We will evaluate 42 patients, all men, with established atherosclerotic disease. Patients will be evaluated in a crossed manner: each subject receives both treatments, intervention and control (in random order), and they will be divided into 2 groups: A and B. In the first intervention stage, after 2 weeks of washout for all patients , group A receives Red Wine (RW) and group B is the control, abstemious. In the 2nd stage of intervention, after 2 weeks of washout for all patients the groups are inverted: group B receives RW; and group A will be abstemious. In the period with wine intervention, patients will receive 250 mL/day of red wine per day, for 5 days of the week, for 3 weeks. Patients will maintain their usual diet without the use of prebiotics or probiotics, or other polyphenolic derivatives. At the beginning and at the end of each stage, patients will be submitted to serum TMAO and intestinal microbiota evaluation. For the intestinal microbiota evaluation, the new generation sequencing will be used in the highly preserved portion of the 16S subunit of the rRNA gene. The determination of TMAO in plasma will be by liquid chromatography coupled to mass spectrometry. Expected results: It is expected to determine if RW acts on the intestinal flora to the point of influencing plasma TMAO concentration.

ELIGIBILITY:
Inclusion Criteria:

1. Men, 45-70 years
2. Established atherosclerotic diseases defined as:

A. Previous history of CAD: angina or acute myocardial infarction (AMI), myocardial revascularization or angioplasty, angiographic evidence of stenosis ≥50% in at least one of the major coronary arteries B. Cerebrovascular disease: transient ischemic stroke or cerebrovascular accident C. Peripheral arterial disease: clinical evidence of extracoronary atherosclerosis

Exclusion Criteria:

1. Acute events in the last 30 days (AMI, troponin elevation, coronary angioplasty or coronary artery bypass grafting)
2. Heart Failure (NYHA functional class ≥ II)
3. Renal Failure (clearance creatinine <30 mL / min by the Cockcroft-Gault formula)
4. Hepatic Failure
5. Gastro-intestinal cancer
6. Intestinal inflammatory diseases
7. Obstructive biliary diseases
8. Prior gastrointestinal surgeries: cholecystectomy or colectomy
9. Use of antibiotics within the last 2 months or during protocol
10. Alcoholism or alcohol intolerance
11. Diabetes mellitus or use of antidiabetics drugs

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 42 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
Gut flora modification assessed by 16S ribosomal rNA gene sequencing and plasma concentration of TMAO changes measured by liquid chromatography coupled to mass spectrometry in 42 patients after ingestion 250 mL of Red Wine 5 days/week, for 3 weeks | up to 10 weeks
  Patients will be divided into 2 groups: A and B. In the first intervention stage, after 2 weeks of washout for all patients , group A receives Red Wine (RW) and group B is the control, abstemious. In the 2nd stage of intervention, after 2 weeks of washout for all patients the groups are inverted: group B receives RW; and group A will be abstemious. In the period with wine intervention, patients will receive 250 mL/day of red wine per day, for 5 days of the week, for 3 weeks. Patients will maintain their usual diet without the use of prebiotics or probiotics, or other polyphenolic derivatives. At the beginning and at the end of each stage, patients will be submitted to serum TMAO and intestinal microbiota evaluation. For the intestinal microbiota evaluation, the new generation sequencing will be used in the highly preserved portion of the 16S subunit of the rRNA gene. The determination of TMAO in plasma will be by liquid chromatography coupled to mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Protasio L da Luz, Professor, Study Chair — Instituto do Coração - InCor - University of Sao Paulo General Hospital; Elisa A Haas, MD, Principal Investigator — Instituto do Coração - InCor - University of Sao Paulo General Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tang WH, Wang Z, Levison BS, Koeth RA, Britt EB, Fu X, Wu Y, Hazen SL. Intestinal microbial metabolism of phosphatidylcholine and cardiovascular risk. N Engl J Med. 2013 Apr 25;368(17):1575-84. doi: 10.1056/NEJMoa1109400. PMID 23614584
- [Background] Zoetendal EG, Collier CT, Koike S, Mackie RI, Gaskins HR. Molecular ecological analysis of the gastrointestinal microbiota: a review. J Nutr. 2004 Feb;134(2):465-72. doi: 10.1093/jn/134.2.465. PMID 14747690
- [Background] Eckburg PB, Bik EM, Bernstein CN, Purdom E, Dethlefsen L, Sargent M, Gill SR, Nelson KE, Relman DA. Diversity of the human intestinal microbial flora. Science. 2005 Jun 10;308(5728):1635-8. doi: 10.1126/science.1110591. Epub 2005 Apr 14. PMID 15831718
- [Background] Andersson AF, Lindberg M, Jakobsson H, Backhed F, Nyren P, Engstrand L. Comparative analysis of human gut microbiota by barcoded pyrosequencing. PLoS One. 2008 Jul 30;3(7):e2836. doi: 10.1371/journal.pone.0002836. PMID 18665274
- [Background] Brown JM, Hazen SL. The gut microbial endocrine organ: bacterially derived signals driving cardiometabolic diseases. Annu Rev Med. 2015;66:343-59. doi: 10.1146/annurev-med-060513-093205. PMID 25587655
- [Background] Ridaura VK, Faith JJ, Rey FE, Cheng J, Duncan AE, Kau AL, Griffin NW, Lombard V, Henrissat B, Bain JR, Muehlbauer MJ, Ilkayeva O, Semenkovich CF, Funai K, Hayashi DK, Lyle BJ, Martini MC, Ursell LK, Clemente JC, Van Treuren W, Walters WA, Knight R, Newgard CB, Heath AC, Gordon JI. Gut microbiota from twins discordant for obesity modulate metabolism in mice. Science. 2013 Sep 6;341(6150):1241214. doi: 10.1126/science.1241214. PMID 24009397
- [Background] Caricilli AM, Saad MJ. The role of gut microbiota on insulin resistance. Nutrients. 2013 Mar 12;5(3):829-51. doi: 10.3390/nu5030829. PMID 23482058
- [Derived] Haas EA, Saad MJA, Santos A, Vitulo N, Lemos WJF, Martins AMA, Picossi CRC, Favarato D, Gaspar RS, Magro DO, Libby P, Laurindo FRM, Da Luz PL; WineFlora Study. A red wine intervention does not modify plasma trimethylamine N-oxide but is associated with broad shifts in the plasma metabolome and gut microbiota composition. Am J Clin Nutr. 2022 Dec 19;116(6):1515-1529. doi: 10.1093/ajcn/nqac286. PMID 36205549